CLINICAL TRIAL: NCT05627492
Title: Pragmatic Patient-oriented Extension Study of Dialectical Behavior Therapy Booster Sessions for Youth With and/or at Familial Risk for Bipolar Disorder
Acronym: DB2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Benjamin Goldstein, Director of the Centre for Youth Bipolar Disorder, Clinician-Scientist, Professor of Psychiatry, Pharmacology & Toxicology, and Psychological Clinical Science, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 099/2022
Record Dates: First submitted 2022-11-17; First posted 2022-11-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Bipolar Disorder
Keywords: Youth; Dialectical Behavior Therapy (DBT); Suicide; Psychotherapy
MeSH Terms: conditions — Bipolar Disorder; Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth with and/or at familial risk for bipolar disorder (Experimental): 120 youth aged 14 to 26 with bipolar disorder (type I, type II, not otherwise specified/NOS via KSADS-PL or SCID-5-RV) OR at high-risk for bipolar disorder (parent or sibling with bipolar disorder type I or II via KSADS-PL or SCID-5-RV) will be enrolled in the dialectical behavioral therapy booster session intervention.
  Interventions: Behavioral: Dialectical behavioral therapy

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy — DBT will be conducted over 2 years. Participants and their treatment providers will decide on the frequency of sessions collaboratively. This may include individual and/or skills sessions in addition to phone coaching for those who attend individual sessions at least once per month. DBT consultation will also remain a component of the treatment. Participants may choose skills training, conducted in approximately 60 minute meetings, and individual therapy conducted in approximately 60 minute sessions. Family participation in skills training is highly encouraged. Skills training may include: psychoeducation, mindfulness skills, emotion regulation skills, distress tolerance skills, interpersonal skills, and walking the middle path skills. Individual therapy sessions aim to aid the youth in applying skills in their daily lives. We adopt the standard DBT hierarchy of treatment targets.
  Other Names: DBT

SUMMARY:
The study intervention is DBT adapted for youth with and/or at familial risk for bipolar disorder. Participants will have completed one full year of DBT in a previous study. This study is examining use of booster sessions. It is delivered in the form of individual sessions and skills sessions, based on the preference of the study participant. The study participant may also receive skills coaching via phone. There is no standard reference therapy/comparator against which the study intervention is being compared.

DETAILED DESCRIPTION:
The study intervention is DBT adapted for youth with and/or at familial risk for bipolar disorder. Participants will have completed one full year of DBT in a previous study. This study is examining use of booster sessions. It is delivered in the form of individual sessions and skills sessions, based on the preference of the study participant. The study participant may also receive skills coaching via phone. DBT consists of four components: individual therapy sessions, skills sessions, skills coaching via phone, and consultation team. Given this study is an extension of an existing study of full DBT, the proposed intervention is not prescriptive; that is, we have opted not to dictate how many sessions participants will receive and/or when. Instead, we have opted to leave this decision for participants and their treatment providers to reach collaboratively. Participants, in consultation with their study therapist, will select the frequency of their booster sessions. This may include individual and/or skills sessions in addition to phone coaching for those who attend individual sessions at least once per month. DBT consultation will also remain a component of the treatment. This level of intervention seems appropriate, given that participants have completed a full year of DBT and thus may require a less intensive treatment for continued care. Moreover, it is important to give youth autonomy in treatment options to model health decision making for other life choices.

ELIGIBILITY:
Inclusion Criteria

The participant must meet all of the inclusion criteria to eligible for this clinical trial:

1. Has completed participation in the DB1 study (049-2021) or the DB3 study (009-2021);
2. English speaking;
3. Age 14 years, 0 months to 26 years, 11 months;
4. Meets diagnostic criteria for bipolar disorder by KSADS-PL(< 20 years of age) OR SCID-5-RV (≥ 20 years of age) OR have a biological parent/sibling with BD (type I or II) confirmed via KSADS-PL or SCID-5-RV;
5. Followed by a psychiatrist who provides ongoing care;
6. If BD-I, taking ≥1 mood stabilizing medication (i.e., antimanic anticonvulsant, antipsychotic, and/or lithium);
7. Able and willing to give informed consent/assent to participate.

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this clinical trial:

1. A life-threatening medical condition requiring immediate treatment;
2. Current victim of sexual or physical abuse;
3. Current substance use disorder other than mild cannabis or alcohol use disorder;
4. Evidence of mental retardation, moderate to severe autism spectrum disorder, or organic central nervous system disorder by the K-SADS-PL, parent report, medical history, or school records that would interfere with active participation in DBT.

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Total number of DBT sessions used during the study interval measured using the Therapy Tracking Form | At the end of study completion (five years)
  The Therapy Tracking Form will be used to document the date of the therapy session, type of session, session duration, content, and scheduled date for next therapy visit. This form will be completed by the study therapist after each therapy session.
Number of unscheduled/expedited DBT sessions that are required measured using the Therapy | At the end of study completion (five years)
  The Therapy Tracking Form will be used to document if the session was a scheduled session or an unscheduled/expedited session. This form will be completed by the study therapist after each therapy session.
Frequencies of different factors/circumstances leading to the need for unscheduled/expedited DBT sessions measured using the Therapy | At the end of study completion (five years)
  The Therapy Tracking Form will be used to document the reason for the unscheduled/expedited DBT session. This form will be completed by the study therapist after each therapy session.

SECONDARY OUTCOMES:
Adherence score for DBT booster sessions measured using a modified version of the Dialectical Behavior Therapy Adherence Checklist - Individual Therapy | At the end of study completion (five years)
  Video recordings will be rated for adherence using a modified version of the Dialectical Behavior Therapy Adherence Checklist - Individual Therapy (DBT AC-I) [54]. The 12 DBT strategy domains will be rated as yes/no: 1) structural strategies; 2) problem assessment strategies; 3) problem solving strategies; 4) contingency management strategies; 5) exposure strategies; 6) cognitive modification strategies; 7) validation strategies; 8) reciprocal communication strategies; 9) irreverent communication strategies; 10) dialectical strategies; 11) case management strategies; 12) protocols.
Frequencies of specific DBT components (individual sessions, skills session, phone coaching) measured using the Therapy Tracking Form | At the end of study completion (five years)
  The Therapy Tracking Form will be used to document the type of therapy session and phone coaching use. This form will be completed by the study therapist after each therapy session.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 12 months to 18 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 18 months to 24 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SID-P uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 12 months to 15 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 15 months to 18 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 18 months to 21 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 21 months to 24 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 12 months to 18 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 18 months to 24 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 12 months to 18 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 18 months to 24 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 12 months to 15 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 15 months to 18 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 18 months to 21 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 21 months to 24 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Treatment Satisfaction Questionnaire (18-item) | 15 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 18 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 21 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 24 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 12 months to 15 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 15 months to 18 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 18 months to 21 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 21 months to 24 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 12 months to 15 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 15 months to 18 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 18 months to 21 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 21 months to 24 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 24 months to 30 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SIDP uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in symptoms using the Structured Interview for DSM-IV Personality Disorders (SIDP-IV): Borderline Personality Disorder | 30 months to 36 months
  Borderline and antisocial personality symptoms will be assessed using the Structured Interview for DSM-IV Personality. The SIDP uses a semi structured interview format to assess for symptoms of personality disorders. Scores one each item range from 0 to 3 and high scores indicate symptoms of borderline personality disorder and levels of impairment.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 24 months to 27 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 27 months to 30 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 30 months to 33 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in suicidality using the Suicidal Ideation Questionnaire (SIQ) | 33 months to 36 months
  Youth participants will complete the self-report Suicidal Ideation (SIQ), which is intended to identify participants whose level of suicidal ideation is severe enough to warrant further intervention. Each item is rated on a 7-point Likert-type scale (0= "I never had this thought" to 6="almost every day") and is used to indicate the frequency with which the participant experiences each thought.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 24 months to 30 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in symptoms using the Adolescent Longitudinal Interval Follow-up Evaluation (ALIFE) | 30 months to 36 months
  The Longitudinal Interval Follow-up Evaluation (LIFE) will provide a comprehensive cross-sectional and longitudinal picture of the symptomatic and psychosocial course and outcome of all participants in this study. Scores range from 0-3 on certain disorders and 0-6 for other disorders. High scores indicate high level of symptom impairment.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 24 months to 30 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS) | 30 months to 36 months
  Suicidal events (past and over follow-up) will be assessed with the Pediatric Version of the Columbia-Suicide Severity Rating Scale (C-SSRS). The C-SSRS has sound psychometric properties, yields ratings of widely accepted definitions of youth suicidal events, and was used in other pediatric treatment trials yielding standardized outcomes to compare across studies. This is a semi-structured interview that includes yes/no questions as well as narrative. It captures number of suicidal events as well as type and severity.
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 24 months to 27 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 27 months to 30 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 30 months to 33 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Change in emotion regulation using the Difficulties in Emotion Regulation Scale (DERS) | 33 months to 36 months
  Youth participants will complete the Difficulties in Emotion Regulation (DERS), a 36-item questionnaire assessing emotional dysregulation. Participants indicate how often each item applies to them on a scale from 1="almost never; 0-10 percent" to 5= "almost always; 91-100 percent".
Treatment Satisfaction Questionnaire (18-item) | 24 months to 27 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 27 months to 30 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 30 months to 33 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Treatment Satisfaction Questionnaire (18-item) | 33 months to 36 months
  During follow-up visits, participants, parents, and/or siblings who are participating in therapy sessions will complete an 18-item Treatment Satisfaction Questionnaire. This assesses clients' satisfaction of the service (responses range from quite dissatisfied to very satisfied) as well as whether or not the service addressed the clients' needs.
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 24 months to 27 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 27 months to 30 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 30 months to 33 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in use of DBT skills with the DBT Ways of Coping Checklist (DBT-WCCL) | 33 months to 36 months
  Youth participants will complete the DBT-WCCL, a 59-item questionnaire assessing the use of DBT skills and coping strategies. Participants indicate how often they engaged in the thought/behavior from 0= "never used" to 3= "regularly used".
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 24 months to 27 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 27 months to 30 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 30 months to 33 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.
Change in temperament using the Conflict Behavior Questionnaire (CBQ) | 33 months to 36 months
  The Conflict Behavior Questionnaire (CBQ) is a youth and parent 20-item self-report instrument that taps into conflict and negative communication between parents and their children. Items are rated as "true" or "false". Higher scores indicate greater levels of conflict and negative communication.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada